CLINICAL TRIAL: NCT05240040
Title: Radioembolization to Treat Primary and Metastatic Liver Tumors
Brief Title: Treat Primary and Metastatic Liver Tumors
Status: Withdrawn | Type: Observational
Why Stopped: Resources
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 029.HPB.2016.D
Record Dates: First submitted 2019-04-03; First posted 2022-02-15 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2022-02

CONDITIONS: Intrahepatic Cholangiocarcinoma; Liver Tumor; Metastatic Cancer; Metastatic Liver Cancer
Keywords: Intrarterial glass; Radiospheres; Liver Cancer; Intrahepatic
MeSH Terms: conditions — Cholangiocarcinoma; Carcinoma, Hepatocellular; Neoplasm Metastasis; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The use of Radiospheres in the management of intrahepatic cholangiocarcinoma is largely unknown and not reported in the medical literature. Methodist Dallas Medical Center has a large volume of IR procedures with Radioembolization and the investigators feel it is imperative to understand the outcomes, risks and benefits of the therapy in order to formulate recommendation to other centers.

DETAILED DESCRIPTION:
A retrospective chart review of patients who have the diagnosis of intrahepatic cholangiocarcinoma. Only patients treated at MDMC are included and data will be obtained from Meditech and Epic. A non-identified database of cases with the diagnosis of intrahepatic cholangiocarcinoma already treated with radiospheres will be created and compared with cases treated by other means.

Intrahepatic cholangiocarcinoma is the second most common primary malignancy of the liver. The standard therapy has been resection but many cases are not resectable due to comorbidities or other poor surgical candidacy factors. Most of these patients end up getting chemotherapy which can be toxic and sometimes poorly tolerated. Intrarterial glass or resin radioembolization has been used and published from only 3 centers in the medical literature and it has been shown to be a reasonable alternative to the above options. At MDMC, this therapy has been used effectively and it is important to describe the investigator's experience.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of intrahepatic cholangiocarcinoma from January 2006 until April 2017 at Methodist Dallas Medical Center (MDMC)
* Patients 18 years old or older

Exclusion Criteria:

* Patients without the diagnosis of intrahepatic cholangiocarcinoma
* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have the diagnosis of intrahepatic cholangiocarcinoma and were treated at MDMC .
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
review the outcomes of patients treated with radiospheres | January 2006 until April 2017
  Patient survival
time to recurrence | January 2006 until April 2017
  time to recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Mejia, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States